CLINICAL TRIAL: NCT04967573
Title: Prophylactic vs Therapeutic Anticoagulation in Symptomatic Isolated Distal Deep Vein Thrombosis (IDENT): a Prospective, Multicenter, Single-blind, Randomized Controlled Trial
Brief Title: Prophylactic vs Therapeutic Anticoagulation in Symptomatic Isolated Distal Deep Vein Thrombosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2021-175R
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Anticoagulation (Experimental): Rivaroxaban 10 mg od for 3 months
  Interventions: Drug: Rivaroxaban
- Therapeutic Anticoagulation (Active Comparator): Rivaroxaban 20 mg od for 3 months
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 20 mg or 10 mg for 3 months

SUMMARY:
The efficacy and safety of anticoagulant treatment is not established for patients with acute symptomatic isolated distal deep vein thrombosis (IDDVT). The latest Antithrombotic Therapy for VTE Disease Guideline suggested using the same anticoagulation as for patients with acute proximal DVT in patients with acute IDDVT. However, a single-center retrospective cohort study found therapeutic anticoagulation was associated with an increase risk of bleeding. Thus, this study aimed to assess the short-term risk of recurrent venous thrombotic events and bleeding events in patients with a first acute symptomatic IDDVT of the leg treated with prophylactic or therapeutic anticoagulant therapy with rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90
* Outpatients with a first, acute (within 2 weeks), symptomatic, objectively confirmed isolated distal DVT
* Compliance to the scheduled follow up plan
* Ability and willing to participate and sign the informed consent.

Exclusion Criteria:

* Any absolute contraindication to anticoagulant treatment
* Pregnancy or breast-feeding
* Systolic pressure > 180 mmHg or diastolic pressure > 100 mmHg
* Platelet count < 100 × 10⁹ /L
* Serum creatinine > 180 mmol/L or creatinine clearance ≤30 ml/min
* Liver disease associated with coagulopathy and high risk of bleeding
* Clinically suspected or confirmed pulmonary embolism
* Ipsilateral or contralateral proximal DVT
* Any indication for long-term anticoagulation
* Enrolled in another clinical trial simultaneously
* Life expectancy < 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographically confirmed recurrent venous thromboembolism | 6 months
  Recurrent venous thromboembolism includes proximal extension of isolated distal DVT, new contralateral proximal DVT and pulmonary embolism.
Major or clinically relevant non-major bleeding events | 3 months
  Major bleeding events are defined according to the International Society on Thrombosis and Haemostasis criteria. Clinically relevant non-major bleeding events refer to which do not meet the mentioned criteria of major bleeding but need at least an unscheduled in-person consultant.

SECONDARY OUTCOMES:
Individual component of primary outcomes (e.g. proximal extension, major bleeding) | 6 months
  Individual component of primary outcomes, including proximal extension of isolated distal DVT, new contralateral proximal DVT, new pulmonary embolism, major bleeding events, clinically relevant non-major bleeding events.
Residual vein occlusion | 6 months
Post-thrombotic syndrome | 6 months
All-cause death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Shi, PhD, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Huadong Hospital affiliated to Fudan University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Wusong Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou M, Zhang W, Zhang Y, Xie T, Mao J, Shi Z. Therapeutic or prophylactic anticoagulation in acute isolated distal deep vein thrombosis: protocol for a prospective, multicentre, single-blind, randomised controlled trial (TOP-IDDVT). BMJ Open. 2022 Feb 28;12(2):e056826. doi: 10.1136/bmjopen-2021-056826. PMID 35228291